CLINICAL TRIAL: NCT04903015
Title: Cerebral and Cognitive Modifications in Retired Professional Soccer Players as Compared to Non Exposed to Repeated Cranial Impacts Sportsmen : Transverse Analytic Study
Brief Title: Cerebral and Cognitive Impact of Professional Soccer Practice
Acronym: TC-FOOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 8077
Record Dates: First submitted 2021-05-10; First posted 2021-05-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Chronic Encephalopathy
Keywords: traumatic chronic encephalopathy; soccer; MRI; neuropsychology; head traumatism
MeSH Terms: conditions — Chronic Traumatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- professional Soccer players (Experimental)
  Interventions: Diagnostic Test: MRI
- athletes not exposed to head injuries. (Active Comparator)
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — The following sequences of the MRI will be acquired during the inclusion visit:
  * 3D T1 gradient echo (GRE): anatomy; registration; cerebral, white matter, and grey matter volumetry; and cortical thickness;
  * multiecho 3D T2 GRE: quantitative susceptibility mapping (QSM), iron overload quantification;
  * continuous arterial spin labeling (ASL) 3D: cerebral perfusion;
  * resting-state fMRI: functional connectivity;
  * 64-direction DTI (b=1000 and 2500): alterations in white matter and its microstructure, anatomic connectivity;
  * monovoxel spectroscopy of the mesencephalus with short echo time (TE).

SUMMARY:
The objective of this study is to evaluate, using MRI, the microstructural consequences and the onset of any cognitive impairment in professional soccer players at the end of their career, who have experienced repeated minor head injuries. Over the long term, these head injuries could lead to morphological lesions and have an impact on soccer players' cognitive skills.

The main evaluation criterion corresponds to the modifications found on MRI in the professional soccer player group (diffusion tensor, cerebral perfusion, fMRI, cerebral volumetry and cortical thickness, spectroscopy, susceptibility imaging).

This is an exposure/nonexposure study assessing the onset of MRI abnormalities (diffusion tensor, cerebral perfusion, fMRI, volumetry and cortical thickness, spectroscopy, susceptibility imaging) in professional soccer players exposed to repeated mild head injuries, who are either at the end of their career or retired for approximately 10 years, compared to high-level athletes not exposed to head injuries.

ELIGIBILITY:
Inclusion Criteria:

Exposed high-level athletes: professional soccer players at the end of their career (32- years old) playing in France Ligue 1 or 2 exposed to repeated mild head injuries with no history of severe head injury or cerebral lesion;

-High-level athletes not exposed to repeated mild head injuries: control group paired for age with professional soccer players, who have never regularly participated in sports exposing them to head injuries (notably rugby, basketball, handball, American football, hockey, combat sports, etc.) and who have no history of head injury, even mild. Professional tennis players or former players will be preferentially recruited.

Exclusion Criteria:

* Refusal to participate in the study;
* refusal to be informed of abnormalities on MRI
* Incapacity to give informed consent or under a legal protection order;
* History of cerebral concussion including the presence after head shock of one or more of the following signs or symptoms: a period of confusion or disorientation, a period of loss of consciousness of 30 minutes or less, post-traumatic amnesia not exceeding 24 hours
* History of severe head/brain injury;
* History of neurological or psychiatric disorder;
* Known cerebral abnormality diagnosed by an imaging exam (CT or MRI);
* History or regular or occasional consumption of drugs, unweaned active smoking or weaned for less than 1 year, excessive consumption of alcohol (> 20 g alcohol per day, evaluated with the formula "degree of alcohol × volume in cl × 8/1000"), weaned or not.
* Usage of medication targeting the central nervous system in the 2 weeks preceding inclusion in the study;
* Prior history of severe hypertension, diabetes, chronic heart disease, progressive or disabling disease;
* Contraindication to MRI (claustrophobia, implanted material not compatible with MRI, refusal to be informed of abnormality discovered on MRI);

Ages: 32 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Abnormalities on MRI in professional soccer players exposed to repeated mild head injuries, potentially related to chronic traumatic encephalopathy, compared to high-level athletes who are not exposed to head injuries. | day 1
  This is a study assessing the relation between exposure to mild head injuries during soccer play in professional players and the onset of MRI and neuropsychological abnormalities. The main evaluation criterion corresponds to the quantitative MRI modifications (professional soccer player group compared with control group).

SECONDARY OUTCOMES:
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  RL RI 16 items (Van der Linden, 2001) to assess the functioning of verbal episodic memory (= 25 min.)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Memory reproduction of Rey's complex figure in order to assess episodic visual memory (Rey Osterrieth, 1941) (= 20 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Verbal and visuo-spatial auditory empans (Wechsler scale Memory form III, 1997) to assess short-term memory and working memory (= 5 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Copy of Rey's complex figure (Rey-Osterrieth, 1941) assessing visual-constructive abilities and planning (= 5 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  The Brixton Test, a spatial anticipation task that also evaluates executive functioning (Burgess P.W. & Shallice T. (1996) (= 15 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Trail Making Test A and B (Reitan et al., 1950) assessing treatment speed and mental flexibility (= 5 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Computerized attention tests will also be used to measure reaction times and also executive aspects (Phasic Alert, Split Attention and Zimmermann APR Incompatibility version 2.1, 2009) (= 15 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Social cognition test Reading the Mind in the eyes assessing the ability to read the emotions of others which, in turn, is related to pSocial cognition test Reading the Mind in the eyes assessing the ability to read the emotions of others which, in turn, is related to performance in team problem-solving tasks (Baron-Cohen; 2001) ( = 10 min)
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  A BRIEF-A (Behavioural Evaluation Inventory of Executive Functions - Adult Version): 10min
The cognitive impact of repeated mild head injuries via a neuropsychological evaluation by neurophysiological tests: number of errors and time to complete tests | day 1
  Research into recurrent symptoms such as headache (seniority, frequency), fatigability, sleep disturbance, dizziness, blurred vision, photo-phonophobia

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane KREMER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Kepka S, Lersy F, Godet J, Blanc F, Bilger M, Botzung A, Kleitz C, Merignac J, Ohrant E, Garnier F, Pietra F, Noblet V, Deck C, Willinger R, Kremer S. Cerebral and cognitive modifications in retired professional soccer players: TC-FOOT protocol, a transverse analytical study. BMJ Open. 2022 Nov 9;12(11):e060459. doi: 10.1136/bmjopen-2021-060459. PMID 36351716